CLINICAL TRIAL: NCT06900803
Title: Pharmacist-Led Education Through Interactive Visualization Dashboards for Adherence Support and Sustained Involvement in Sacubitril/Valsartan Therapy for Patients With Heart Failure With Reduced Ejection Fraction (PharmD ASSIST HFrEF): Study Protocol for Implementation in a Parallel-Group, Pragmatic Randomized Controlled Trial
Brief Title: Evaluating Dashboard-Integrated Pharmacist-Led Education on Improving Sacubitril/Valsartan Adherence in Heart Failure (PharmD ASSIST HFrEF)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202501197RINC
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HFrEF); Sacubitril/Valsartan; Medication Adherence
Keywords: heart failure with reduced ejection fraction; medication adherence; dashboard; health information technology; patient education; pharmacist; pragmatic trial; randomized controlled trial; sacubitril/valsartan; implementation
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low Adherence Cluster - Intervention Group (Experimental): Dashboard interventions integrated into pharmacist-led education in the low adherence cluster
  Interventions: Device: interactive visualization dashboard (the Enhancing Sacubitril/valsartan Adherence from Initiation to Continuation [ESAIC] dashboard)
- Low Adherence Cluster - Control Group (No Intervention): Pragmatic pharmacist-led education, without dashboard interventions, in the low adherence cluster
- High Adherence Cluster - Intervention Group (Experimental): Dashboard interventions integrated into pharmacist-led education in the high adherence cluster
  Interventions: Device: interactive visualization dashboard (the Enhancing Sacubitril/valsartan Adherence from Initiation to Continuation [ESAIC] dashboard)
- High Adherence Cluster - Control Group (No Intervention): Pragmatic pharmacist-led education, without dashboard interventions, in the high adherence cluster

INTERVENTIONS:
Device: interactive visualization dashboard (the Enhancing Sacubitril/valsartan Adherence from Initiation to Continuation [ESAIC] dashboard) — The dashboard serves as an interactive communication tool during education sessions, promoting real-time dialogue between patients and pharmacists. By collaboratively entering patient-specific data, patients gain insight into personalized visual representations of actionable risk factors. Initially, data specific to the patient are inputted to generate a baseline assessment, presenting hazard ratios that indicate the current condition and pinpoint areas needing improvement. To simulate potential changes, an alternative dataset is deliberately entered, portraying either improvement or deterioration in the patient's status, thereby acting as a motivational tool. Throughout the education session, the dashboard continuously updates hazard ratios, enabling direct comparisons of patient outcomes under varying conditions or treatment scenarios. This dynamic process clearly demonstrates individualized risk-benefit trade-offs in diverse treatment contexts.
  Arms: High Adherence Cluster - Intervention Group; Low Adherence Cluster - Intervention Group

SUMMARY:
The goal of this pragmatic clinical trial is to evaluate whether pharmacist-led education, integrated with interactive visualization dashboards, can enhance medication adherence in patients with heart failure who are prescribed sacubitril/valsartan. The main question it aims to answer is: Can pharmacist-led interactive visualization dashboards improve adherence to sacubitril/valsartan compared to usual care without the dashboard intervention?

Researchers will compare patients receiving pharmacist-led education with interactive dashboards to those receiving standard education, assessing differences in medication adherence and clinical outcomes, among others.

Participants will:

* Complete baseline and follow-up questionnaires on medication adherence and satisfaction with pharmacist-provided services, and others.
* Engage in education sessions led by pharmacists, with or without dashboard integration.

The study outcomes will include medication adherence, and secondary outcomes such as patient satisfaction with pharmacist-provided services, optimized guideline-directed medical therapy score, time to high medication adherence, the calculated proportion of days covered, New York Heart Association functional classification, and the net promoter score used for evaluating recommendation and satisfaction with the dashboard intervention.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 20 or older
* a diagnosis of HFrEF, which is defined by a left ventricular ejection fraction of 40% or less
* currently receiving sacubitril/valsartan at the time of recruitment
* receiving care at the cardiology department or cardiology ward at National Taiwan University Hospital
* referral from the clinicians at National Taiwan University Hospital

Exclusion Criteria:

* unable or unwilling to provide informed consent, adhere to study protocols, or complete required questionnaires in person during three scheduled visits (i.e., 3, 6, 12 months after the baseline measurement)
* having received care at the pharmacist-led HF clinic at National Taiwan University Hospital

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-07 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Medication adherence to sacubitril/valsartan | From enrollment to the end of treatment at 12 months (four key time points: baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3) post-randomization).
  Medication adherence will be assessed using the Morisky 8-item Medication Adherence Scale (MMAS-8) for sacubitril/valsartan, with scores ranging from 0 to 8, where higher scores indicate better medication adherence.

SECONDARY OUTCOMES:
Patient satisfaction with pharmacist-provided services | From enrollment to the end of treatment at 12 months (four key time points: baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3) post-randomization).
  Patient satisfaction will be assessed using the adapted Traditional Chinese version of the modified Patient Satisfaction with Pharmacist Services Questionnaire 2.0 (C-mPSPSQ 2.0). C-mPSPSQ 2.0 is a 6-item scale, with scores ranging from 4 to 24, where higher scores indicate better patient satisfaction with pharmacist-provided services.
Optimized guideline-directed medical therapy (GDMT) score | From enrollment to the end of treatment at 12 months (four key time points: baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3) post-randomization).
  The score, adapted from the ΔGDMT score from Man et al. (2024) and the Optimization Potential Score from Verma et al. (2023), is calculated by dividing the received dose by the target dose based on each class of GDMT according to the current HF guidelines, ranging from 0 to 1 per medication of GDMT. The maximum total score per patient is 5, with four pillars of GDMT and extra one point for a switch from ACEI/angiotensin receptor blockers to sacubitril/valsartan due to the complexity of reimbursement in Taiwan. If valid reasons for not prescribing GDMT are documented in the electronic health records, a score of 1 will still be assigned for each instance.
Medication adherence to guideline-directed medical therapy (GDMT) | From enrollment to the end of treatment at 12 months (four key time points: baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3) post-randomization).
  Medication adherence will be assessed using the Morisky 8-item Medication Adherence Scale (MMAS-8) for GDMT, with scores ranging from 0 to 8, where higher scores indicate better medication adherence.
Time to high medication adherence | From enrollment to the end of treatment at 12 months (four key time points: baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3) post-randomization).
  The time to achieving high medication adherence (defined as a score of 8 on the Morisky 8-item Medication Adherence Scale [MMAS-8]) will be analyzed separately for patients who attain high adherence to sacubitril/valsartan and guideline-directed medical therapy (GDMT), with scores ranging from 0 to 8, where higher scores indicate better medication adherence.
Proportion of days covered (PDC) | From enrollment to the end of treatment at 12 months (four key time points: baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3) post-randomization).
  The PDC will also be calculated to triangulate and validate the results of the Morisky 8-item Medication Adherence Scale (MMAS-8). The data of the PDC will be accessed through the National Health Insurance MediCloud System in Taiwan. The PDC for each guideline-directed medical therapy (GDMT) is calculated by the total days covered in the period divided by the total prescription days in the period, with the common threshold of 80% indicating acceptable medication adherence.
New York Heart Association (NYHA) functional classification | From enrollment to the end of treatment at 12 months (four key time points: baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3) post-randomization).
  The NYHA functional classification, which categorizes heart failure severity into four classes based on symptoms and limitations to physical activity, will be assessed by pharmacists.
Net Promoter Score (NPS) | From enrollment to the end of treatment at 12 months (two key time points: baseline (T0) and 3 months (T1) post-randomization).
  The level of participant endorsement for the intervention (i.e., the ESAIC dashboard) will help identify areas for further enhancement and support its integration into routine clinical practice. The NPS ranges from 1 to 10, with increments of 1, and is classified into three distinct categories: promoters (scoring 9 or 10), passives (scoring 7 or 8), and detractors (scoring 6 or below). In this trial, both pharmacists and patients will provide NPS ratings.

IPD SHARING:
Plan to Share IPD: No
We believe that safeguarding patient confidentiality is of utmost importance, and the current study protocol does not include provisions for public data sharing.